CLINICAL TRIAL: NCT03349658
Title: Evaluation of the Effects of Spinal Versus General Anesthesia on Transcranial Cerebral Oxygen Saturation in Geriatric Patients Undergoing Total Hip Arthroplasty
Brief Title: Cerebral Oximetry and Anesthetic Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AntalyaTRH 17
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Disorder of Hip Joint
Keywords: total hip arthroplasty; cerebral oxygen saturation; general anesthesia; spinal anesthesia
MeSH Terms: interventions — Anesthesia, General; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- general anesthesia (Active Comparator): Patients in this group were randomized to receive general anesthesia.
  Interventions: Other: general anesthesia
- spinal anesthesia (Active Comparator): Patients in this group were randomized to receive spinal anesthesia.
  Interventions: Other: spinal anesthesia

INTERVENTIONS:
Other: general anesthesia — effect of general anesthesia on transcranial regional cerebral oxygen saturation
  Arms: general anesthesia
Other: spinal anesthesia — effect of spinal anesthesia on transcranial regional cerebral oxygen saturation
  Arms: spinal anesthesia

SUMMARY:
The purpose of the study is to compare the effects of spinal and general anesthesia on transcranial regional cerebral oxygen saturation in geriatric patients undergoing total hip arthroplasty.

DETAILED DESCRIPTION:
Geriatric patients who received anesthesia undergoing total hip arthroplasty were randomized by means of a computer-generated randomization order into two groups; general anesthesia group (Group 1) and spinal anesthesia group (Group 2). Before and after induction of the general or spinal anesthesia, patients were monitorized with near infrared spectroscopy for regional cerebral oxygen saturation. Findings were compared statistically.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo elective total hip arthroplasty
* American Society of Anesthesiologists class 1 to 3
* Ability to consent

Exclusion Criteria:

* Pulmonary disease
* History of allergic reaction to local anaesthetics
* Peripheral neuropathy
* Neurologic disease
* Coagulation disorders

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in transcranial regional cerebral oxygenation (rSO2) | 60 minutes
  Assessed every 5 minutes during the procedure

SECONDARY OUTCOMES:
Post anesthetic complications | 1 day
  During stay at the post anesthetic care unit. Any new neurological symptoms etc

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Dagdelen, MD, Study Director — Antalya Training and Research Hospital; Nilgun Kavrut Ozturk, MD, Principal Investigator — Antalya Training and Research Hospital; Ali Sait Kavakli, MD, Principal Investigator — Antalya Training and Research Hospital; Ülkü Arslan, MD, Principal Investigator — Antalya Training and Research Hospital